CLINICAL TRIAL: NCT03612115
Title: Investigation of the Effects of Neuromuscular Electrical Stimulation in Patients With Pulmonary Arterial Hypertension
Brief Title: Neuromuscular Electrical Stimulation in Pulmonary Arterial Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Buse Ozcan Kahraman, Principal Investigator, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2217-GOA
Record Dates: First submitted 2018-07-27; First posted 2018-08-02 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neuromuscular electrical stimulation intervention (Experimental): Neuromuscular electrical stimulation treatment
  Interventions: Device: Neuromuscular electrical stimulation
- Control (No Intervention): No additional intervention

INTERVENTIONS:
Device: Neuromuscular electrical stimulation — Neuromuscular electrical stimulation to the bilateral deltoid and quadriceps femoris muscles with 50 Hz for 3 days/week, 8 weeks.
  Device name: Four-channel Wireless Professional (DJO United Kingdom Ltd., Chattanooga, France)
  Arms: Neuromuscular electrical stimulation intervention

SUMMARY:
This study aimed to investigate the effects of neuromuscular electrical stimulation on peripheral muscles and other physical and psychosocial variables in patients with pulmonary arterial hypertension. This study was designed as an assessor-blind randomized controlled trial. Thirty-one patients with pulmonary arterial hypertension will be recruited. The participants will randomly divided two parallel groups as treatment and control. For the treatment group, neuromuscular electrical stimulation will be applied to the bilateral deltoid and quadriceps femoris muscles with 50 Hz for 3 days/week, 8 weeks. Control group will not be received any additional treatment, just given healthy life recommendations such as walking. The participants will be assessed before and after the treatment by a blind assessor to the group allocation. The outcome measure will be assessments of the upper and lower limb muscle strength, respiratory muscle strength, muscle cross-sectional area and thickness, pulse wave velocity, exercise capacity, walking speed, functional mobility and balance performances, balance confidence, fatigue perceptions, physical activity level, activities of daily living and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Elevated pulmonary artery pressures measured by right heart catheterization
* New York Heart Association class II or III
* Stabile Pulmonary Arterial Hypertension-specific pharmaceutical therapy for 3 months

Exclusion Criteria:

* Orthopaedic problems
* Significant restrictive or obstructive pulmonary disease
* Acute cor pulmonale.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-09-28 (Actual); Study Completion 2017-09-28 (Actual)

PRIMARY OUTCOMES:
Isometric muscle strength | Change from Baseline at 8 weeks
  Isometric muscle strength for knee extensors

SECONDARY OUTCOMES:
Isometric muscle strength | Change from Baseline at 8 weeks
  Isometric muscle strength for shoulder flexors and abductors
Hand grip strength | Change from Baseline at 8 weeks
  Hand grip strength
Quadriceps femoris muscle thickness | Change from Baseline at 8 weeks
Rectus femoris cross-sectional area | Change from Baseline at 8 weeks
Pulse wave velocity | Change from Baseline at 8 weeks
Six-Minute Walk Test | Change from Baseline at 8 weeks
Six-Minute Pegboard and Ring Test | Change from Baseline at 8 weeks
Sit-to-Stand Test | Change from Baseline at 8 weeks
Timed-Up and Go Test | Change from Baseline at 8 weeks
Activities-specific Balance Confidence Scale | Change from Baseline at 8 weeks
  The Activities-specific Balance Confidence Scale is a 16-item instrument designed to measure a patient's perceived level of confidence in performing common activities of daily living without losing balance and falling. The patient ranks his confidence to complete each item from 0% (no confidence) to 100% (complete confidence). Total score is calculated as sum score ranged from 0 to 100. Higher scores indicate higher balance confidence level.
4-m Gait Speed Test | Change from Baseline at 8 weeks
Fatigue Impact Scale | Change from Baseline at 8 weeks
  The Fatigue Impact Scale is widely used to measure fatigue. It is a 40-item multidimensional scale measuring the physical, cognitive and social. Patients are asked to rate how much of a problem fatigue has caused them during the past month, including the day of testing, on a 5-point Likert-type scale, with response options ranging from 0 "no problem" to 4 "extreme problem". Higher scores indicate the greater level of fatigue (total score ranged from 0 to 160).
International Physical Activity Questionnaire-Short Form | Change from Baseline at 8 weeks
  The International Physical Activity Questionnaire-Short Form has 7 items listing activities and requests estimates of durations and frequencies for each activity engaged in over the past week. Durations are multiplied by known metabolic equivalents per activity and the results for all items are summed for the overall physical activity score. Scores for walking and for moderate and vigorous activities are sums of corresponding item scores. Higher scores indicate higher physical activity level.
Milliken Activities of Daily Living Scale | Change from Baseline at 8 weeks
  Milliken Activities of Daily Living Scale consists of 47 items including preparing meals, and eating (8 items), self-care (9 items), dressing oneself (8 items), manual manipulation of objects (9 items), house cleaning, and washing clothes (7 items), and other activities (6 items). For scoring the level of ability to perform each item, a 5-point scale, and for the level of necessity to perform these items, a 3-point scale is used. Total score can range from 0 to 705 points. Higher scores indicate less limitation in activities of daily living.
Nottingham Health Profile | Change from Baseline at 8 weeks
  Health-related quality of life will be assessed using Nottingham Health Profile scale which is a general quality of life questionnaire that measures perceived health problems and their impact on normal daily activities. It has 38 items divided into six domains: energy level, pain, emotional reactions, sleep, social isolation and physical abilities. Items use yes/no answer format and each item is weighted. Total scores for each domain range from 0 to 100. Higher scores represent less quality of life in relevant domain.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylül University, Izmir, Turkey (Türkiye)